CLINICAL TRIAL: NCT06447389
Title: "Clinical Evaluation of Retraction Cord Effectiveness Using Direct Digitalization Method in Determining the Preparation Margin Line"
Brief Title: "Clinical Evaluation of Retraction Cord Effectiveness Using Intraoral Scanner
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Kıvanç Akça, Prof. Dr., Hacettepe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: KA-22056
Record Dates: First submitted 2024-06-02; First posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Prosthesis User; Digitalism
Keywords: digital dentistry; effectiveness; retraction cord

STUDY DESIGN:
Masking Description: The investigator, who performed the statistical analysis, will not know which group the obtained primary and secondary data belong to until all evaluations are completed.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evaluation of the Effectiveness of Retraction Cord (Other): For each case, two tooth-supported restorations will be produced: one with and one without the application of a retraction cord. The accuracy of the marginal fit of the produced restorations will be determined through digital analysis of the data.
  Interventions: Other: retraction cordu (SURE-CORD®PLUS)

INTERVENTIONS:
Other: retraction cordu (SURE-CORD®PLUS) — The evaluation of the effectiveness of retraction cords in determining the restoration margin in the fabrication of short fixed partial dentures for patients with missing teeth.

SUMMARY:
Dental-supported fixed partial dentures (FPDs) have long been a commonly preferred treatment method for the rehabilitation of teeth with excessive substance loss and for addressing existing tooth deficiencies. Crucial factor affecting the success and quality of FPDs is the marginal fit of the restoration. Marginal discrepancy refers to the vertical or horizontal gap between the restoration finish line and the preparation finish line. To achieve high marginal fit restorations, gingival retraction techniques are used with the aim of removing the marginal gingiva away from the finish line. Retraction cords are commonly used for this purpose nowadays. The aim of the study is to evaluate the effect of retraction cords on the preparation finish line and the marginal fit of produced restorations using direct digital measurement methods.

DETAILED DESCRIPTION:
This study is designed to produce temporary bridges based on two supporting teeth, fabricated using an intraoral scanner, and to evaluate the marginal fit of these bridges based on two different digital measurements obtained with and without the use of retraction cord on the patient.

The study will encompass patients with a single missing tooth in the posterior region of the lower or upper jaw, specifically involving the second premolar or first molar, planned for a three-unit tooth-supported fixed partial denture (SPP). Prior to preparation, patients will be examined for the assessment of the soft tissue around the teeth, and data collection will be conducted in accordance with the criteria outlined in Table-1, following the guidelines of the 2017 Consensus Report on the Classification of Periodontal and Peri-implant Diseases and Conditions regarding periodontal health and gingival diseases in healthy and reduced periodontium.

Subsequently, the abutment teeth will be prepared stepwise using high-speed rotary instruments and diamond preparation burs to accommodate fixed restorations.

The study groups will be formed considering the presence or absence of retraction application. The groups will be defined as Group I (No retraction cord) and Group II (Retraction cord present).

In Group I, digital impressions will be taken directly in all patients without placing a retraction cord.

In Group II, digital impressions will be taken in the same patients using a "000" knitted retraction cord and a single retraction cord technique.

As part of this plan, digital impressions of the abutment teeth for the temporary bridge will be taken both before and after the application of the retraction cord. The temporary bridges fabricated from these impressions will then be evaluated intraorally.

For each case included in the study, the .stl files from the initial impression for the restoration, the post-production impression, and the restoration itself will be superimposed and digitally analyzed using reverse engineering software.

The depths of the preparation finish lines will be recorded using a probe. The recorded depths of the preparation finish lines and the amounts of marginal discrepancy of the restorations will be examined together. Based on the obtained data, the effect of the preparation finish line depth on the marginal fit of the restorations will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation after reading and understanding the informed consent form.
* Over 18 years of age with no general health issues.
* Presence of a single missing posterior tooth in the upper or lower jaw.
* Possession of "clinical gingival health" in terms of periodontal condition ("Clinical gingival health of a healthy periodontium is defined as the absence of bleeding on probing, erythema, edema, symptoms, and no loss of bone or attachment.(17))
* Teeth with less than half of the tooth structure lost that do not require post-core treatment.

Exclusion Criteria:

* Failure to accept voluntary participation in the study after reading the informed consent form.
* General health condition being unsuitable for prosthetic treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
Digital analysis | 1.5 year
  The comparison of the marginal fit of restorations fabricated from digital data with and without the use of a retraction cord was performed using reverse engineering software. The digital scans taken after preparation, the digital scans taken after restoration delivery, and the .stl files of the restorations were superimposed within the software and analyzed for marginal fit.

SECONDARY OUTCOMES:
Probing dept | 1.5 year
  Secondary data will be collected by measuring the step depths on the abutment teeth after preparation. These measurement points will be compared with the marginal fit of the temporary bridges at the same points, and the effect of step depth on marginal fit will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Kıvanç Akça, DDS,PhD, Principal Investigator — Hacettepe University Faculty of Dentistry Department of Prosthodontics Ankara, Turkey
Locations (1):
- Hacettepe University Faculty of Dentistry Department of Prosthodontics, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Acar O, Erkut S, Ozcelik TB, Ozdemir E, Akcil M. A clinical comparison of cordless and conventional displacement systems regarding clinical performance and impression quality. J Prosthet Dent. 2014 May;111(5):388-94. doi: 10.1016/j.prosdent.2013.08.009. Epub 2013 Dec 18. PMID 24360008
- [Result] Martins FV, Santana RB, Fonseca EM. Efficacy of conventional cord versus cordless techniques for gingival displacement: A systematic review and meta-analysis. J Prosthet Dent. 2021 Jan;125(1):46-55. doi: 10.1016/j.prosdent.2019.09.009. Epub 2020 Jan 31. PMID 32008797
- [Result] Mangano FG, Margiani B, Solop I, Latuta N, Admakin O. An Experimental Strategy for Capturing the Margins of Prepared Single Teeth with an Intraoral Scanner: A Prospective Clinical Study on 30 Patients. Int J Environ Res Public Health. 2020 Jan 7;17(2):392. doi: 10.3390/ijerph17020392. PMID 31936096
- [Result] Huang C, Somar M, Li K, Mohadeb JVN. Efficiency of Cordless Versus Cord Techniques of Gingival Retraction: A Systematic Review. J Prosthodont. 2017 Apr;26(3):177-185. doi: 10.1111/jopr.12352. Epub 2015 Sep 17. PMID 26378615